CLINICAL TRIAL: NCT02000622
Title: A Phase III, Open Label, Randomised, Controlled, Multi-centre Study to Assess the Efficacy and Safety of Olaparib Monotherapy Versus Physicians Choice Chemotherapy in the Treatment of Metastatic Breast Cancer Patients With Germline BRCA1/2 Mutations.
Brief Title: Assessment of the Efficacy and Safety of Olaparib Monotherapy Versus Physicians Choice Chemotherapy in the Treatment of Metastatic Breast Cancer Patients With Germline BRCA1/2 Mutations.
Acronym: OlympiAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0819C00003; 2013-005137-20 (EudraCT Number)
Record Dates: First submitted 2013-11-18; First posted 2013-12-04 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Metastatic; BRCA 1 Gene Mutation; BRCA 2 Gene Mutation
Keywords: Breast Cancer; Metastatic; Olaparib; BRCA; PARP inhibitor; HER2; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olaparib (Experimental): Olaparib tablet 300mg bd po
  Interventions: Drug: Olaparib
- Physician's choice chemotherapy (Active Comparator): Capecitabine 2500 mg/m2 d1-14 q 21, or Vinorelbine 30 mg/m2 d1,8 q 21, or Eribulin 1.4 mg/m2 d1,8 q 21
  Interventions: Drug: Physician's choice chemotherapy

INTERVENTIONS:
Drug: Olaparib — Patients will be administered olaparib orally twice daily (bid) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water.
  Arms: Olaparib
Drug: Physician's choice chemotherapy — Investigators will declare one of the following regimens:
  * Capecitabine 2500 mg/m2 po daily (divided in 2 doses) x 14 days, repeat every 21 days
  * Vinorelbine 30 mg/m2 IV Day 1 and Day 8, repeat every 21 days
  * Eribulin 1.4 mg/m2 IV Day 1 and Day 8, repeat every 21 days
  Arms: Physician's choice chemotherapy

SUMMARY:
This open label, randomised, controlled, multi-centre phase III study will assess the efficacy and safety of single agent olaparib vs standard of care based on physician's choice of capecitabine, vinorelbine or eribulin in metastatic breast cancer patients with gBRCA 1/2 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious.
* Histologically or cytologically confirmed breast cancer with evidence of metastatic disease.
* Prior therapy with an anthracycline and a taxane in either an adjuvant or metastatic setting.
* Prior platinum allowed as long as no breast cancer progression occurred on treatment or if given in adjuvant/neoadjuvant setting at least 12 months from last dose to study entry elapsed.
* ER/PR breast cancer positive patients must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy.
* ECOG performance status 0-1.
* Adequate bone marrow, kidney and liver function.

Exclusion Criteria:

* Prior treatment with PARP inhibitor.
* Patients with HER2 positive disease.
* More than 2 prior lines of chemotherapy for metastatic breast cancer.
* Untreated and/or uncontrolled brain metastases.
* Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry. Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix, DCIS or stage I grade 1 endometrial cancer allowed.
* Known HIV (Human Immunodeficiency Virus) infection.
* Pregnant or breast-feeding women.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center, New York
Locations (136):
- United States (38):
  - Research Site, San Diego, California
  - Research Site, Santa Rosa, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Plantation, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Lafayette, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, Commack, New York
  - Research Site, Harrison, New York
  - Research Site, New York, New York
  - Research Site, Rockville Centre, New York
  - Research Site, Syracuse, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Germantown, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Burlington, Vermont
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- China (12):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
- Czechia (3):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- France (5):
  - Research Site, Caen
  - Research Site, Montpellier
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Villejuif
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Nyíregyháza
  - Research Site, Veszprém
- Italy (5):
  - Research Site, Bologna
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (8):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kagoshima
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Suita
- Mexico (4):
  - Research Site, Estado de México
  - Research Site, Mérida
  - Research Site, México
  - Research Site, San Juan del Río
- Peru (3):
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, San Borja
- Poland (6):
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Grzepnica
  - Research Site, Lodz
  - Research Site, Tarnobrzeg
  - Research Site, Warsaw
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Russia (7):
  - Research Site, Arkhangelsk
  - Research Site, Ivanovo
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Saransk
  - Research Site, Yaroslavl
- South Korea (5):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Oviedo
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Zurich
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (9):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Konya
  - Research Site, Mersin
- United Kingdom (6):
  - Research Site, Aberdeen
  - Research Site, Colchester
  - Research Site, Coventry
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, Delaloge S, Li W, Tung N, Armstrong A, Wu W, Goessl C, Runswick S, Conte P. Olaparib for Metastatic Breast Cancer in Patients with a Germline BRCA Mutation. N Engl J Med. 2017 Aug 10;377(6):523-533. doi: 10.1056/NEJMoa1706450. Epub 2017 Jun 4. PMID 28578601
- See also: Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1910&filename=D0819C00003_Clinical_Study_Protocol_Final_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 27 March 2014 and the last patient on 30 October 2015. Patients were randomized at 125 centres across 19 countries in North America, South America, Europe and Asia.
Pre-assignment Details: Screening occurred in 2 parts. Part 1: patients with unknown BRCA status were tested by Myriad. Part 1 screening failures were mostly due to no BRCA1/2 mutation detected. Part 2: patients with a known germline BRCA mutation were screened. 302 patients were randomized.
Period: Overall Study
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Started | 205 | 97
Completed | 36 | 17
Not Completed | 169 | 80
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 4 | 0
Not completed — Death | 159 | 73
Not completed — Withdrawn due to site closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set consisting of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300 mg bd | Chemotherapy | Total
Number analyzed (Participants) | 205 | 97 | 302
Age, Continuous [Median (Full Range); unit: Years]
  Age (years) | 44 [22 to 76] | 45 [24 to 68] | 44 [22 to 76]
Age, Customized [Count of Participants; unit: Participants]
  <50 | 138 | 63 | 201
  >=50-<65 | 56 | 30 | 86
  >=65 | 11 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 95 | 295
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 66 | 28 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 134 | 63 | 197
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Global: BULGARIA | 4 | 4 | 8
  Global: CHINA | 32 | 9 | 41
  Global: CZECH REPUBLIC | 11 | 1 | 12
  Global: FRANCE | 5 | 4 | 9
  Global: HUNGARY | 10 | 0 | 10
  Global: ITALY | 17 | 7 | 24
  Global: JAPAN | 15 | 9 | 24
  Global: KOREA | 11 | 9 | 20
  Global: MEXICO | 1 | 4 | 5
  Global: PERU | 3 | 1 | 4
  Global: POLAND | 10 | 5 | 15
  Global: ROMANIA | 1 | 1 | 2
  Global: RUSSIAN FEDERATION | 10 | 5 | 15
  Global: SPAIN | 7 | 6 | 13
  Global: SWITZERLAND | 6 | 2 | 8
  Global: TAIWAN | 1 | 1 | 2
  Global: TURKEY | 8 | 6 | 14
  Global: UNITED KINGDOM | 8 | 4 | 12
  Global: UNITED STATES | 45 | 19 | 64
Receptor status [Count of Participants; unit: Participants] — ER = oestrogen receptor, PgR = progesterone receptor. All patients were HER2 negative.
  Participants
    ER and/or PgR positive | 103 | 49 | 152
    ER and PgR negative | 102 | 48 | 150
Received prior chemotherapy for metastatic breast cancer [Count of Participants; unit: Participants]
  Yes | 146 | 69 | 215
  No | 59 | 28 | 87
Received prior platinum for breast cancer [Count of Participants; unit: Participants]
  Yes | 60 | 26 | 86
  No | 145 | 71 | 216

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Using Blinded Independent Central Review (BICR) According to Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1)
Description: Time from randomisation to the earliest of objective radiological progression or death by any cause in the absence of objective progression. Objective radiological progression is defined using Response Evaluation Criteria In Solid Tumours (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Radiological scans performed at baseline then every ~6 weeks up to 24 weeks, then every ~ 12 weeks thereafter until objective radiological disease progression. Assessed up to a maximum of 30 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Olaparib 300 mg bd: Olaparib 300 mg bd tablets
- Chemotherapy: Physician's choice of chemotherapy; capecitabine, vinorelbine, or eribulin
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 7.0 [5.7 to 8.3] | 4.2 [2.8 to 4.3]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Study is sized to provide 90% power to detect a true treatment effect of PFS hazard ratio 0.653; Test type: Superiority; p = 0.0009, Log Rank — A priori threshold for statistical significance (2-sided) is 0.05; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.43 to 0.80] — Hazard ratio <1 favours olaparib

2. Secondary Outcome: Time to Second Progression or Death (PFS2)
Description: Time from randomisation to the earliest of the progression event subsequent to the first objective radiological progression, or death. Second progression may involve any of; objective radiological or symptomatic progression or death. Objective radiological progression is defined using Response Evaluation Criteria In Solid Tumours (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Symptomatic progression is assessed by investigators based on clinical examination.
Time Frame: Second progression status reviewed every 8 weeks following the first objective radiological progression as per investigator assessment. Assessed up to a maximum of 30 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 13.2 [10.9 to 15.3] | 9.3 [7.3 to 10.4]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Test type: Superiority; p = 0.0033, Log Rank — PFS2 tested using a multiple testing procedure with a recycling strategy. With 157 PFS2 events, a priori threshold for statistical significance (2-sided) was 0.008; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.40 to 0.83] — Hazard ratio <1 favours olaparib

3. Secondary Outcome: Overall Survival (OS)
Description: Time from randomisation until death due to any cause.
Time Frame: Survival status reviewed every 3 weeks until treatment discontinued, then every 8 weeks. Assessed up to a maximum of 30 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 19.3 [16.7 to 21.8] | 19.6 [14.1 to 24.2]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Test type: Superiority; p = 0.5665, Log Rank — OS tested using a multiple testing procedure with a recycling strategy. With 140 OS events, a priori threshold for statistical significance (2-sided) was 0.018; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.63 to 1.29] — Hazard ratio <1 favours olaparib

4. Secondary Outcome: Objective Response Rate (ORR) Using Blinded Independent Central Review (BICR) Data Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1)
Description: Number of responders according to blinded independent central review (BICR) assessment. Per Response Evaluation Criteria In Solid Tumours Criteria (RECIST v1.1) for target lesions assessed by CT or MRI: Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions; Overall Response = CR + PR.
Time Frame: as for outcome 1
Population: Evaluable For Response (EFR) Analysis Set consisting of all randomised patients with measurable disease at baseline, i.e. at least one measurable target lesion assessed by blinded independent central review (BICR)
Measure: Number; unit: Participants
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 167 | 66
Participants | 100 | 19

5. Secondary Outcome: Adjusted Mean Change in Global Health Status/Quality of Life (QoL) Score From the European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Change from baseline in global health status/quality of life (QoL) score assessed using a mixed model for repeated measures (MMRM) analysis, including all post-baseline global health status/QoL scores up to the latest scheduled visit where at least 20 patients on each treatment arm have a score. Global health status/QoL score is on a scale from 0 to 100. A higher score represents an improved health status/QoL.
Time Frame: EORTC QLQ-C30 assessments performed at baseline then every ~6 weeks until objective radiological disease progression. Assessed up to a maximum of 30 months.
Population: Subset of Full Analysis Set (FAS) consisting of all randomised patients with an evaluable baseline EORTC QLQ-C30 assessment and at least one evaluable post-baseline assessment
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 191 | 73
Score on a scale | 3.9 [1.5 to 6.3] | -3.6 [-8.0 to 0.8]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Test type: Superiority; p = 0.0035, Mixed Models Analysis; Variables for treatment, visit, treatment-visit interaction, adjusted for baseline global health status/QoL score, baseline score-visit interaction; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [2.5 to 12.4] — Mean difference >0 favours olaparib

6. Secondary Outcome: Progression-free Survival (PFS) Using Blinded Independent Central Review (BICR) According to Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) in Patients Confirmed as Myriad CDx gBRCAm
Description: Time from randomisation to the earliest of objective radiological progression or death by any cause in the absence of objective progression. Objective radiological progression is defined using Response Evaluation Criteria In Solid Tumours Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Assessed in patients with a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (gene sequencing and large rearrangement analysis).
Time Frame: as for outcome 1
Population: Subset of Full Analysis Set (FAS) consisting of all randomised patients who were confirmed as Myriad CDx gBRCAm
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 202 | 95
Months | 7.4 [5.7 to 8.3] | 4.2 [2.8 to 4.3]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Test type: Superiority; p = 0.0005, Log Rank; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.41 to 0.78] — Hazard ratio <1 favours olaparib

7. Other Pre Specified Outcome: Time to First Subsequent Cancer Therapy or Death (TFST)
Description: Time from randomisation to the earliest of first subsequent cancer therapy start date following study treatment discontinuation, or death.
Time Frame: Subsequent cancer therapy status reviewed every 8 weeks following study treatment discontinuation. Assessed up to a maximum of 30 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 9.4 [8.3 to 10.6] | 4.2 [3.3 to 5.2]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Supportive analysis to PFS; Test type: Superiority; p < 0.0001, Log Rank; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.24 to 0.47] — Hazard ratio <1 favours olaparib

8. Other Pre Specified Outcome: Time to Second Subsequent Cancer Therapy or Death (TSST)
Description: Time from randomisation to the earliest of second subsequent cancer therapy start date following study treatment discontinuation, or death.
Time Frame: as for outcome 7
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 14.3 [12.2 to 15.5] | 10.5 [8.4 to 11.3]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Supportive analysis to PFS2; Test type: Superiority; p = 0.0002, Log Rank; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.38 to 0.74] — Hazard ratio <1 favours olaparib

9. Secondary Outcome: Overall Survival (OS) at Final OS
Description: Time from randomisation until death due to any cause.
Time Frame: Survival status reviewed every 3 weeks until treatment discontinued, then every 8 weeks. Assessed up to a maximum of 40 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 19.3 [17.2 to 21.6] | 17.1 [13.9 to 21.9]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Test type: Superiority; p = 0.5131, Log Rank — OS tested using a multiple testing procedure with a recycling strategy. With 192 OS events, a priori threshold for statistical significance was 0.045; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.66 to 1.23] — Hazard ratio <1 favours olaparib

10. Secondary Outcome: Overall Survival (OS) at Extended OS
Description: Time from randomisation until death due to any cause.
Time Frame: Survival status reviewed every 3 weeks until treatment discontinued, then every 8 weeks until Sep 2017 (final OS DCO), then every 3 months. Assessed up to a maximum of 64 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 19.3 [17.2 to 21.6] | 17.1 [13.9 to 21.9]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Test type: Superiority; p = 0.4167, Log Rank; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.67 to 1.18] — Hazard ratio <1 favours olaparib

11. Other Pre Specified Outcome: Time to First Subsequent Cancer Therapy or Death (TFST) at Extended OS
Description: as for outcome 7
Time Frame: Subsequent cancer therapy status reviewed every 8 weeks following study treatment discontinuation until Sep 2017 (final OS DCO), then every 3 months. Assessed up to a maximum of 64 months.
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 9.4 [8.3 to 10.6] | 4.3 [3.4 to 5.4]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Supportive analysis to PFS; Test type: Superiority; p < 0.0001, Log Rank; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.27 to 0.50] — Hazard ratio <1 favours olaparib

12. Other Pre Specified Outcome: Time to Second Subsequent Cancer Therapy or Death (TSST) at Extended OS
Description: as for outcome 8
Time Frame: as for outcome 11
Population: Full Analysis Set (FAS) consisting of all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Chemotherapy
Number analyzed (Participants) | 205 | 97
Months | 14.3 [12.3 to 15.7] | 10.5 [8.5 to 11.3]
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Chemotherapy; Supportive analysis to PFS2; Test type: Superiority; p < 0.0001, Log Rank; Stratified by received prior chemotherapy for metastatic breast cancer (yes/no) and receptor status; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.40 to 0.72] — Hazard ratio <1 favours olaparib

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected throughout the study until study completion (up to a maximum of 30 months). They are reported from date of first dose of study treatment until the earliest of 30 days after last dose of study treatment and data cut-off.
Description: Adverse events and serious adverse events are reported in the Safety Analysis Set including all patients who received at least one dose of study treatment (n=296). Six patients on the chemotherapy arm did not receive any study treatment and therefore are excluded from the Safety Analysis Set, leaving n=91 patients on the chemotherapy arm. All cause mortality is reported in the Full Analysis Set (n=302).
Groups:
- Olaparib 300 mg bd; Chemotherapy: Description (Arm-group)
Arm/Group | Olaparib 300 mg bd | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 159/205 | 73/97
Serious Adverse Events (participants affected / at risk) | 37/205 | 15/91
Other Adverse Events (participants affected / at risk) | 196/205 | 85/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd (N=205) | Chemotherapy (N=91)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 2 (2)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd (N=205) | Chemotherapy (N=91)
Anaemia (Blood and lymphatic system disorders) | 76 (129) | 21 (29)
Leukopenia (Blood and lymphatic system disorders) | 23 (55) | 9 (40)
Lymphopenia (Blood and lymphatic system disorders) | 14 (30) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 37 (89) | 27 (78)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (20) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 14 (16) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 15 (16) | 5 (5)
Constipation (Gastrointestinal disorders) | 26 (30) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 42 (68) | 19 (29)
Dyspepsia (Gastrointestinal disorders) | 17 (20) | 4 (4)
Nausea (Gastrointestinal disorders) | 119 (175) | 31 (40)
Stomatitis (Gastrointestinal disorders) | 16 (23) | 10 (10)
Vomiting (Gastrointestinal disorders) | 66 (127) | 13 (18)
Asthenia (General disorders) | 19 (28) | 12 (15)
Fatigue (General disorders) | 61 (80) | 22 (23)
Mucosal inflammation (General disorders) | 5 (5) | 6 (7)
Pyrexia (General disorders) | 27 (35) | 16 (20)
Influenza (Infections and infestations) | 14 (15) | 4 (4)
Nasopharyngitis (Infections and infestations) | 17 (26) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 27 (40) | 9 (16)
Urinary tract infection (Infections and infestations) | 13 (14) | 3 (3)
Alanine aminotransferase increased (Investigations) | 24 (39) | 16 (19)
Aspartate aminotransferase increased (Investigations) | 20 (29) | 15 (19)
Gamma-glutamyltransferase increased (Investigations) | 13 (14) | 5 (5)
Neutrophil count decreased (Investigations) | 21 (49) | 17 (43)
Platelet count decreased (Investigations) | 10 (19) | 6 (10)
White blood cell count decreased (Investigations) | 33 (75) | 19 (40)
Decreased appetite (Metabolism and nutrition disorders) | 35 (41) | 11 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (27) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (32) | 8 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (19) | 3 (3)
Dizziness (Nervous system disorders) | 18 (18) | 7 (8)
Dysgeusia (Nervous system disorders) | 17 (22) | 6 (6)
Headache (Nervous system disorders) | 41 (51) | 14 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 9 (10)
Insomnia (Psychiatric disorders) | 13 (14) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (40) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 9 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 12 (13)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 19 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days